CLINICAL TRIAL: NCT03096860
Title: Effect of Concurrent Hookah and Alcohol Consumption on Smoking Topography and Toxicant Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Eleanor Leavens, Principal Investigator, Oklahoma State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NIH/NIDA F31 DA04252
Record Dates: First submitted 2017-03-20; First posted 2017-03-30 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Use, Unspecified; Hookah Smoking
MeSH Terms: conditions — Alcohol Drinking; Water Pipe Smoking | interventions — Exercise; Ethanol; Economics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol consumption and hookah (Experimental)
  Interventions: Other: Active alcohol consumption
- Placebo consumption and hookah (Placebo Comparator)
  Interventions: Other: Placebo consumption

INTERVENTIONS:
Other: Active alcohol consumption — Comparison of alcohol consumption vs. placebo consumption and hookah smoking.
  Arms: Alcohol consumption and hookah
Other: Placebo consumption — Comparison of alcohol consumption vs. placebo consumption and hookah smoking.
  Arms: Placebo consumption and hookah

SUMMARY:
The purpose of the current study is to investigate in a prospective randomized cross-over trial, the impact of alcohol versus a placebo drink on smoking behavior and topography (duration and frequency of puffing), abuse liability, and toxicity. It is hypothesized that drinking alcohol before smoking will be associated with longer puffs and shorter duration between puffs and greater abuse liability and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Report using hookah at least 1 time per month over the past 6 months
2. Are at least 21 years old
3. Speak and understand English
4. Do not currently suffer from lung disease including asthma, CF, or COPD
5. Do not currently suffer from heart disease
6. Are not currently pregnant or breast-feeding or have plans to become pregnant or begin breast-feeding at any point during the study
7. No current, regular use of >5 cigarettes or other tobacco products (e.g., e-cig, cigar, etc.) per month.
8. No current marijuana use > 5 times per month
9. No use of illicit drugs during the past 30 days
10. willing to provide informed consent and abstain from all tobacco, nicotine, and marijuana use for at least 12 hours and abstain from alcohol for at least 24 hours prior to each of the two sessions
11. Live within 25 miles of the study location.
12. Have a friend who is eligible and willing to participate.
13. Consume 2 or more or one or more drinks per episode for men and women, respectively
14. Drink alcohol at least one time per week
15. Not currently be seeking treatment for alcohol use
16. Able to answer at least two hookah-specific screening questions from the screener.

    -

Exclusion Criteria:

1. Hookah use less than one time per month over the past 6 months
2. Under the age of 21
3. Unwilling to abstain from alcohol for 24 hours and tobacco and nicotine products 12 hours prior to each study visit
4. Live more than 25 miles from the study location
5. Pregnant or breast feeding or plan to become pregnant or begin breast feeding at any point in the study -

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Total volume smoke inhaled | up to 2 hours
  hookah topography

CONTACTS AND LOCATIONS:
Locations (1):
- The Oklahoma Tobacco Research Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Leavens ELS, Morgan TL, Brett EI, Patzkowsky K, Son J, Molina N, Eissenberg T, Shihadeh A, Leffingwell TR, Wagener TL. Concurrent Alcohol Use and Waterpipe Tobacco Smoking: Smoking Topography, Toxicant Exposure, and Abuse Liability. Nicotine Tob Res. 2020 Feb 6;22(2):280-287. doi: 10.1093/ntr/ntz032. PMID 30820567